CLINICAL TRIAL: NCT06378502
Title: The Effect of Different Antibiotic Protocols for Dental Implant Surgery on Peri-implant Tissue Health and on Oral Microbiome and Resistome
Brief Title: The Effect of Different Antibiotic Protocols on Peri-implant Tissue Health
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Maria Menini, Prof, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: antibiotic-resistence
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-span therapy (Experimental): 1 g Amoxicillin every 8 h starting 1 day before surgery and for 5 days after surgery
  Interventions: Drug: Amoxicillin Long
- Short-span therapy (Experimental): 2 g Amoxicillin 1 h before surgery
  Interventions: Drug: Amoxicillin Short

INTERVENTIONS:
Drug: Amoxicillin Short — Short Span
  Arms: Short-span therapy
Drug: Amoxicillin Long — Long span
  Arms: Long-span therapy

SUMMARY:
The aim of the present project (non-inferiority trial) is to evaluate the effect of different antibiotic strategies (long-span vs. short-span) for implant surgery on peri-implant tissue health, oral microbiome (included resistome) and salivary MiRNomics in healthy patients.

DETAILED DESCRIPTION:
A total of 80 patients will be included and randomly divided in two groups:

1. Long-span prescription: 1 g Amoxicillin every 8 h starting 1 day before surgery and for 5 days after surgery
2. Short-span prescription: 2 g Amoxicillin 1 h before surgery Before surgery, patients will undergo an antibiotic sensitivity test (AST), and non-invasive samples will be taken to analyse oral microbiome including resistome. Saliva samples will be also taken for miRNomics analysis. Patients will be rehabilitated with single implants or partial implant-supported fixed prostheses. The day of surgery, samples of peripheral blood will be taken and peripheral blood mononuclear cells (PBMCs) isolated from the first 30 patients in order to implement a micro-fluidic bioreactor replicating the bone healing process of each patient. 3D bone models will be developed that are suitable for drug screening.

At 2 and 6 months post-treatment, AST test and oral microbiome and resistome analysis will be performed again. 2 months after treatment, a new saliva sample of the patients will be also taken, analysed and compared using MiRnomics technology with the preoperative one with the further aim of identifying reliable biomarkers of mucositis and perimplantitis. During the 12-month follow-up implant survival rate, marginal bone loss (MBL), biologic and technical complication rate and peri-implant health parameters (including plaque index, probing depth and bleeding on probing) will be evaluated.

Parametric or non-parametric comparative tests, as appropriate, will be performed to detect differences between the groups in the various outcome variables. The effect of patient-related and implant-related predictive factors on the various outcomes will be evaluated using multilevel logistic regression analysis. Metadata will be analyzed also with 4th generation Artificial Neural Networks (ANNs) (machine learning) using unsupervised and supervised systems.

Expected results: The present project is expected to clarify if the short-span antibiotic therapy is not inferior to the long-span one in healthy patients undergoing implant surgery. The outcomes will contribute to the development of effective clinical guidelines that will help to tackle the issue of antimicrobial resistance. In addition, the development and validation of a 3D bone model to be used for drug screening is expected, that might overcome limitations of currently available 2D bone models and animal studies. A further expected result is the identification of biomarkers for diagnosis and prognosis in implant dentistry, through salivary miRNomics that might lead to the development of a non-invasive liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers requiring one single implant or partial implant-supported rehabilitation in an edentulous area of the posterior mandible or maxilla

Exclusion Criteria:

* Patients unable to commit to follow-up
* General contraindications to implant surgery
* Immuno-suppressed/immune-compromised patients
* Patients irradiated in the head and/or neck
* Uncontrolled diabetes
* Pregnancy, childbearing potential, breastfeeding
* Smoking habit
* Untreated periodontal disease (Caton et al, J Clin Periodontol 2018)
* Poor oral hygiene and motivation (plaque index > 20%)
* Addiction to alcohol or drugs
* Psychiatric problems and/or unrealistic expectations
* Patients with an acute infection (abscess) or suppuration in the site intended for implant placement
* Patients treated or under treatment with intravenous amino-bisphosphonates
* Patients referred only for implant placement if the follow-up cannot be done at the treatment center
* Patients participating in other studies, if the present protocol could not be fully adhered to
* Patients with allergy/hypersensitivity to penicillin or drug excipients
* Patients recently treated with antibiotics for other indications

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-03 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean peri-implant bone loss | at 6 and 12 months after prosthesis delivery
  bone loss

SECONDARY OUTCOMES:
Incidence of biological and technical complications at the implant site | 12 months
  complications
implant survival rate | 12 months
  CSR
Antibiotic sensitivity | 1 week before and 2 months and 6 months after implant insertion
  sensitivity
Peri-implant myco-, microbiome and resistome | 1 week before and 2 months and 6 months after implant insertion
  resistome
Salivary miRNomics | 1 week before and 2 months after implant insertion
  miRNomics
Adverse reactions | during the entire follow-up period
  reaction
Development of a 3D bone model | 1 year
  3D bone model
Plaque index (PI) | 3, 6 and 12 months after prosthesis delivery
  measured on 6 surfaces each tooth - percentage value
Bleeding on probing (BOP) | 3, 6 and 12 months after prosthesis delivery
  measured on 6 surfaces each tooth - percentage value
Peri-implant pocket probing depth (PPD) | 3, 6 and 12 months after prosthesis delivery
  measured on 6 surfaces each tooth - percentage value

IPD SHARING:
Plan to Share IPD: Undecided